CLINICAL TRIAL: NCT01432496
Title: A Multicentric, Randomized, Controlled, Double Blinded, Phase III Clinical Trial; Comparing Peritoneal Nebulization of Ropivacaine 150 mg With Peritoneal Nebulization of Saline
Brief Title: Peritoneal Nebulization of Ropivacaine for Pain Control After Laparoscopic Colectomy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: There was insuficient recruitment in two centers
Sponsor: San Gerardo Hospital (Other)
Collaborators: University of Milano Bicocca (Other); Azienda Ospedaliera di Lecco (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); University of Pavia (Other)
Responsible Party: Principal Investigator, Pablo Mauricio Ingelmo M.D., Consultant Anesthesiologys. First Service of Anesthesia and Intensive Care, San Gerardo Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR HSG 06 2010 Colectomy
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Postoperative Pain
Keywords: Laparoscopic; Colectomy; Nebulization; Ropivacaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine 150 mg (Experimental): Nebulization of Ropivacaine 150 mg in the peritoneal cavity with the Aeroneb Pro system
  Interventions: Drug: Ropivacaine 150 mg
- Saline 15 ml (Placebo Comparator): Nebulization of Saline 15 ml in the peritoneal cavity with the Aeroneb Pro system
  Interventions: Drug: saline 15 ml

INTERVENTIONS:
Drug: Ropivacaine 150 mg — Nebulization of Ropivacaine 150 mg in the peritoneal cavity
  Other Names: Nebulization Ropivacaine
  Arms: Ropivacaine 150 mg
Drug: saline 15 ml — Nebulization of saline 15 ml in the peritoneal cavity
  Other Names: Nebulization Saline
  Arms: Saline 15 ml

SUMMARY:
The purpose of this study is to assess if intraperitoneal nebulization of Ropivacaine 150 mg produces better postoperative pain control than Saline nebulization after laparoscopic colectomy.

DETAILED DESCRIPTION:
Recently intraperitoneal nebulization of local anesthetic has been used as an alternative to direct intraperitoneal instillation. Intraperitoneal aerosolization of Bupivacaine 50 mg after laparoscopic cholecystectomy significantly reduced postoperative pain, morphine consumption and incidence of postoperative nausea and vomiting and it is associated with rapid mobilization compared with patients receiving direct instillation of Bupivacaine 50 mg or placebo.

In a recent study the investigators found that nebulization of Ropivacaine 30 mg with the AeronebPro® before or after laparoscopic cholecystectomy and gynecologic laparoscopic surgery reduces postoperative pain and morphine consumption. Patients receiving preoperative nebulization of Ropivacaine presented significantly less postoperative pain (-50% clinical setting) and consumed significant less morphine (-50% and -40% respectively) than patients in control groups during the first 48 hours after surgery.

The effects of peritoneal nebulization of ropivacaine during laparoscopic colectomy on pain control and morphine consumption were not evaluated.

The investigators hypothesize that intraperitoneal nebulization of Ropivacaine may produce better pain control and less morphine consumption than nebulization of saline after laparoscopic colectomy.

ELIGIBILITY:
Inclusion Criteria:

* Females and Males 18-80 years old
* ASA Score I (American Society of Anesthesiologists classification : a normal healthy patient.
* ASA Score II (American Society of Anesthesiologists classification): A patient with mild systemic disease
* ASA Score III (American Society of Anesthesiologists classification): A patient with severe systemic disease
* Patients scheduled for oncological laparoscopic colectomy
* Patients who do not use opioids analgesic drugs before surgery
* Patients without cognitive impairment or mental retardation

Exclusion Criteria:

* Females and Males under 18 or over 80
* ASA Score IV (American Society of Anesthesiologists classification): A patient with severe systemic disease that is a constant threat to life
* ASA Score V (American Society of Anesthesiologists classification): A moribund patient who is not expected to survive without the operation
* Emergency/urgency surgery
* Postoperative admission in an intensive care unit with sedation or ventilatory assistance
* Cognitive impairment or mental retardation
* Use of opiods before surgery
* Progressive degenerative diseases of the CNS
* Convulsions or chronic therapy with antiepileptic drugs
* Severe hepatic or renal impairment
* Allergy to one of the specific drugs under study
* Acute infection or inflammatory chronic disease
* Alcohol or drug addiction
* Any kind of communication problem
* Neurologic or psychiatric disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 72 hours
  Numeric Ranking Scale (NRS 0 to 10 points) at rest (static NRS) and after a deep inspiration or cough (dynamic NRS) in PACU and at 6, 24, 48 and 72 hours after the discharge from PACU.

SECONDARY OUTCOMES:
Time of unassisted walking | 72 hours
  Unassisted walking time is defined as the time in hours between PACU discharge and when the patient is able to walk out of his room and back to bed without any assistance.
Return to active bowel function | 72 hours
  The return of bowel function will be assessed using two parameters: time of first flatus and time of first bowel movement.
Hospital morbidity | 72 hours
  All complications or adverse effects associated or possibly associated with the interventions under study, surgery or anesthesia will be quantified
Time and condition for hospital discharge | 72 hours
  Time in days elapsed between surgery and hospital discharge.
Analgesic consumption | 72 hours
  The total dose of morphine will be quantified using the PACU clinical chart and/or PCA infusers memory display

CONTACTS AND LOCATIONS:
Overall Officials: Pablo M Ingelmo, MD, Principal Investigator — San Gerardo Hospital, MB, Italy
Locations (3):
- Italy (3):
  - Azienda Ospedaliera di Lecco. Presidio "A.Manzoni", Lecco, LC
  - San Gerardo Hospital, Monza, MB
  - Fondazione IRCCS Policlinico San Matteo, Pavia, PV

REFERENCES:
- [Background] Alkhamesi NA, Peck DH, Lomax D, Darzi AW. Intraperitoneal aerosolization of bupivacaine reduces postoperative pain in laparoscopic surgery: a randomized prospective controlled double-blinded clinical trial. Surg Endosc. 2007 Apr;21(4):602-6. doi: 10.1007/s00464-006-9087-6. Epub 2006 Dec 16. PMID 17180268
- [Background] Greib N, Schlotterbeck H, Dow WA, Joshi GP, Geny B, Diemunsch PA. An evaluation of gas humidifying devices as a means of intraperitoneal local anesthetic administration for laparoscopic surgery. Anesth Analg. 2008 Aug;107(2):549-51. doi: 10.1213/ane.0b013e318176fa1c. PMID 18633034
- [Background] Schlotterbeck H, Schaeffer R, Dow WA, Diemunsch P. Cold nebulization used to prevent heat loss during laparoscopic surgery: an experimental study in pigs. Surg Endosc. 2008 Dec;22(12):2616-20. doi: 10.1007/s00464-008-9841-z. Epub 2008 Mar 18. PMID 18347861